CLINICAL TRIAL: NCT00611143
Title: The Effects of Atorvastatin on the Occurrence of Postoperative Atrial Fibrillation After Off-Pump Coronary Artery Bypass Grafting Surgery
Brief Title: Atorvastatin for Prevention of Postoperative Atrial Fibrillation After Off-Pump Coronary Artery Bypass Grafting Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: YK On, MD, PhD / Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006-08-022
Record Dates: First submitted 2008-01-27; First posted 2008-02-08 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Artery Bypass
Keywords: Off-pump coronary artery bypass graft; Atorvastatin; Postoperative atrial fibrillation
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Atorvastatin group
  Interventions: Drug: atorvastatin
- 2 (No Intervention): Control group

INTERVENTIONS:
Drug: atorvastatin — atorvastatin 20 mg/d, started 3 days before surgery
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether pretreatment with atorvastatin protects against atrial fibrillation following off-pump coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
Atrial fibrillation after cardiac surgery is the most common arrhythmic complication that may increase incidence of congestive heart failure, renal insufficiency, and stroke, which increase the length of hospital stay, the rates of re-hospitalization, and cost of care. Its pathogenesis is multifactorial, and its prevention and management remain suboptimal. Recently, observational evidence has suggested that patients who have undergone previous statin therapy have a lower incidence of postoperative atrial fibrillation.

The purpose of this study is to determine whether pretreatment with atorvastatin protects against atrial fibrillation following off-pump coronary artery bypass graft surgery.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients scheduled for the elective off-pump CABG surgery

Exclusion Criteria:

* prior statin use
* previous episodes of atrial fibrillation
* impaired renal function with serum creatinine >2mg/dL
* serum aspartate aminotransferase or alanine aminotransferase concentrations more than 3 times the upper limit of normal
* a malignancy or inflammatory disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2006-05; Primary Completion 2007-04 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
the development of postoperative in-hospital atrial fibrillation confirmed by 12-lead ECG | in-hospital period

SECONDARY OUTCOMES:
major adverse cardiac and cerebrovascular events rate, including cardiovascular death, postoperative stroke, myocardial infarction, or persistent atrial fibrillation,and identification of predictive markers for postoperative atrial fibrillation | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Young Keun On, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Cardiac and Vascular Center; Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Song YB, On YK, Kim JH, Shin DH, Kim JS, Sung J, Lee SH, Kim WS, Lee YT. The effects of atorvastatin on the occurrence of postoperative atrial fibrillation after off-pump coronary artery bypass grafting surgery. Am Heart J. 2008 Aug;156(2):373.e9-16. doi: 10.1016/j.ahj.2008.04.020. Epub 2008 Jun 17. PMID 18657672